CLINICAL TRIAL: NCT06427785
Title: The Effect of Wavelet Index in Monitoring the Sedation Depth of Remimazolam Besylate
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-ke-75
Record Dates: First submitted 2024-04-11; First posted 2024-05-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-04

CONDITIONS: Remimazolam; Anesthesia Awareness; Sedative, Hypnotic, or Anxiolytic Withdrawal
Keywords: Wavelet Index; Remimazolam; Depth of Sedation
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remimazolam group: Thirty patients underwent elective lower extremity surgery receive spinal anesthesia, and then, remimazolam besylate was given intravenously with an induction dose of 3mg/min. When the MOAA/S (Modified Observer's Assessment of Alertness/Sedation) score was ≤1, remimazolam besylate was maintained at 1mg/min for 24min, and finally stopped. Wavelet index, MOAA/S score, blood pressure, heart rate, respiratory rate, and pulse oxygen saturation were continuously monitored during the period.
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Remimazolam besylate — Thirty patients underwent elective lower extremity surgery receive spinal anesthesia, and then remimazolam besylate was given intravenously with an induction dose of 3mg/min. When the MOAA/S (Modified Observer's Assessment of Alertness/Sedation) score was ≤1, remimazolam besylate was maintained at 1mg/min for 24min, and finally stopped. Wavelet index, MOAA/S score, blood pressure, heart rate, respiratory rate, and pulse oxygen saturation were continuously monitored during the period.

SUMMARY:
To explore the sedative effect of remimazolam in patients undergoing spinal anesthesia without pain stimulation. Both the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) and the Wavelet index (WLi) were used to monitor the depth of anesthesia of remimazolam, and exploring the correlation and consistency between MOAA/S score and WLi value at the same time.

DETAILED DESCRIPTION:
Patients undergoing spinal anesthesia were received remimazolam besylate for sedation continuously. Both the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) and the Wavelet index (WLi) were used to monitor the depth of anesthesia of remimazolam, and exploring the correlation and consistency between MOAA/S score and WLi value at the same time.

ELIGIBILITY:
Inclusion Criteria:

* ASA was classified as I-III
* The operation time was less than 120 minutes
* Informed consent is signed by all study participants
* Elective lower extremity surgery under spinal anesthesia was performed

Exclusion Criteria:

* Pregnant or lactating women
* Patients with Difficult Airways
* History of severe neurological and muscular diseases and mental retardation
* Patients with severe respiratory and circulatory diseases, including acute heart failure. Unstable angina pectoris. Resting ECG heart rate <50 beats/min. QTc: ≥470ms in men and ≥480ms in women. Third degree atrioventricular block. Severe arrhythmia. Moderate to severe heart valve disease. Chronic obstructive pulmonary disease. A history of severe asthma.
* Abnormal liver and kidney function: ALT and/or AST exceeding 2.5 times the upper limit of the medical reference range
* Take diazole drugs and/or opioids in one month or nearly three months
* Patients who were allergic to or contraindicated to benzodiazepines, opioids, propofol, flumazenil, naloxone, etc
* Patients who could not monitor the depth of anesthesia for various reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was an unrandomized, single-group study. The sample size was calculated using PASS 15™(NCSS, LLC. Kaysville, Utah, USA.) software. The degree of confidence (1-β) was set at 0.90, and the α value was set at 0.05. ρ0, the baseline correlation, was set to 0. The ρ1, alternating correlation, was set to 0.3 based on the expected minimum r value of 0.3 obtained in previous literature. Final calculations show that 112 pairs of data were needed to complete the experiments. Approximately 20 pairs of data were expected to be recorded per participant, and 30 participants were expected to be enrolled in this study. So, the sample size was adequate.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-08-17 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
The value of the Wavelet index (WLi) when MOAA/S (Modified Observer's Assessment of Alertness/Sedation) score ≤ 1. | Through study completion, an average of 1 day
  Sedation was assessed using the MOAA/S (Modified Observer's Assessment of Alertness/Sedation) scale. It ranges from 5(alert) to 0(deep sedation). Wavelet index (WLi) is a parameter that potentially could be used to regulate the sedative depth of anesthesia. The range of WLi values is 0-100, with a value of 0 indicating no EEG activity, a value of 100 indicating complete wakefulness, and a value of 40-60 taken to indicate an appropriate level of general anesthesia.

SECONDARY OUTCOMES:
Mean time from initiation of drug administration to MOAA/S (Modified Observer's Assessment of Alertness/Sedation) score ≤1 | Through study completion, an average of 1 day
  Sedation was assessed using the MOAA/S (Modified Observer's Assessment of Alertness/Sedation) scale. It ranges from 5(alert) to 0(deep sedation). The mean time from drug administration to MOAA/S score ≤1 was recorded.
The average time from drug withdrawal to full recovery | Through study completion, an average of 1 day
  Sedation was assessed using the MOAA/S (Modified Observer's Assessment of Alertness/Sedation) scale. It ranges from 5(alert) to 0(deep sedation). The mean time from drug withdrawal to MOAA/S score = 5 was recorded